CLINICAL TRIAL: NCT06032429
Title: Effects of the Shared Medical Appointments on Blood Glucose and Self-care Efficacy for Middle-aged Patients With Type 2 Diabetes
Brief Title: Effects of Shared Medical Appointments for Diabetic Patients in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B10703021
Record Dates: First submitted 2021-03-23; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabete Mellitus; Taiwan; effect
MeSH Terms: conditions — Diabetes Mellitus | interventions — Shared Medical Appointments; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Medical Appointments (Experimental): This strategy is conducted by groups of patients meeting over time for comprehensive care, usually involving a practitioner with prescribing privileges, for a defining chronic condition or health care state. Meanwhile, this model often use educational and/or self-management enhancement strategies, paired with medication management, in an effort to achieve improved disease outcomes.
  Interventions: Other: Shared Medical Appointments
- Standard care (No Intervention): Routine health education without more advanced illustration

INTERVENTIONS:
Other: Shared Medical Appointments — SMA is a subset of such clinics and are defined by groups of patients meeting over time for comprehensive care for a defining chronic condition or health care state, which involved both a person trained or skilled in delivering patient education or facilitating patient interaction.
  Other Names: Standard care
  Arms: Shared Medical Appointments

SUMMARY:
This quasi-experimental study is done to investigate the effect of Shared Medical Appointments (SMA) program for the diabetic patients in Taiwan. The relevant corresponding effects were determined via the generalized estimating equation (GEE) model.

DETAILED DESCRIPTION:
Study design and participants A quasi-experimental pre-posttest control group design, with purposive sampling, was used to recruit participants from the Endocrinology department of a hospital in southern Taiwan from Jan to Dec in 2019. The inclusion criteria were (i) being at least 20 years old at the time of recruitment (ii) having no cognitive impairment and severe complications, (iii) being able to express opinions in either Mandarin or Taiwanese, and (iv) having a diagnosis of diabetes. To ensure participants' anonymity, all questionnaires were marked with an encryption code to facilitate data analysis, but with no personal identifiers.

Sample size calculation Sample size calculation for this analysis of repeated measures to detect an effect size of 0.4 at 80% power and a 0.05 significance level indicated that a sample size of 56 patients is needed (according to G- POWER 3.1 analytical software, Franz Faul, Universitat Kiel, Germany). A sample of at least 68 participants for both groups combined was required on the basis of these parameters, allowing for a 20% attrition rate.

Intervention Because continued participation was essential for this study, the participants were divided into the experiment or control group in accordance with the personal willingness. The control group received routine health education lasting for about 30 minutes per medical visit, which consisted of consultation about disease symptoms, related treatments, and self-care skills. They would receive health education instruction leaflets for reference purposes if necessary.

The experiment group received four shared medical appointments (SMP) -based group education sessions (7-10 participants, 1.5 hours each) for four consecutive weeks in addition to routine health education at a private room in the outpatient unit. One registered nurse who received SMP facilitator training, from the Taiwanese Association of Diabetic Educators, served as the class facilitator. SMP sessions were conducted using several colored maps covering different topics, which included "healthy diet and exercises", "relevant treatment towards diabetic medications", " self-monitoring of blood glucose," and "treatment on hypoglycemia and hyperglycemia" . This procedure served to create mutual imagery to be shared with participants. In addition to using these colored maps, the facilitator further offered participants self-designed conversation cards and asked them to share individual glycemic control experiences based on the questions shown on the cards.

Outcome measures The primary outcomes were composed of two self-development tools, namely diabetic self-management questionnaire (DSMQ) as well as diabetic self-care questionnaire (DSCQ).

On the other hand, the consideration of covariates contained additional items addressing demographic and disease characteristics were developed based on clinical experience and literature review, and were collected at study entry via patient interviews and medical records. Demographic data included sex, age, marital status, education level, religion, household status, monthly income, and certain lifestyle factors, such as smoking, exercise habits, and presence of sleep disturbances. Smoking status was recorded as "non-smoker" or "current or ex-smoker." Those who exercised regularly (i.e., weekly) were classified as having "exercise habits." Sleep disturbances were defined as waking up at night more than twice without external factors during the week before the interview. Disease characteristics included the presence of chronic disease (i.e., stroke, hypertension, heart disease, renal disease, or cancer), medication regimen, and duration of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* being at least 20 years old at the time of recruitment,
* having no cognitive impairment and severe complications,
* being able to express opinions in either Mandarin or Taiwanese, and
* having a diagnosis of DM.

Exclusion Criteria:

* being unwillingness to participant this work
* Attending the similar health education program in the past

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the self-management level assessed by the self-developed scale | up to six months

SECONDARY OUTCOMES:
the self-care level assessed by the self-developed scale | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Fan Chen, Study Director — Dalin Tzuchi Hospital, The Buddhist Tzuchi Medical Foundation
Locations (1):
- Pin-Fan Chen, Chiayi City, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided